CLINICAL TRIAL: NCT05445687
Title: Assessment and Rehabilitation of Narrative Language in Children With Hearing Impairment and Developmental Language Disorder
Brief Title: Rehabilitation of Narrative Language in Children With Hearing Impairment and Developmental Language Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sara Magdy Ibrahim, Assistant Lecturer of Phoniatrics, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0201642
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Hearing Impaired Children; Developmental Language Disorder
Keywords: Hearing impairment; Developmental language disorder; Narrative language; Language rehabilitation
MeSH Terms: conditions — Language Development Disorders; Hearing Loss

STUDY DESIGN:
Intervention Model Description: A comparative intervention study comparing the effect of narrative language intervention on narrative language skills in children with hearing impairment and children with developmental language disorder in comparison to conventional language intervention.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcome assessors will be blinded to the type of intervention given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hearing Impairment cases (Experimental): Hearing impaired children who will receive the proposed narrative intervention program.
  The program will include 24 illustrated story sequences with a minimum of 5 sequences representing the main story elements: characters and setting; problems; internal response; actions; and consequence. Story icons will be designed to represent the main 5 elements to accompany storytelling and act as visual prompts.The narrative intervention program will be applied on the cases groups by a phoniatrician in 24 sessions, 60 minutes in duration, one session per week, for 3 months.
  Interventions: Behavioral: Narrative language intervention program
- Hearing Impairment control (Active Comparator): The Hearing impairment control group will receive the conventional language rehabilitation sessions in 30 minute sessions twice a week, for 3 months. Conventional language therapy targets semantics, syntax, prosody, pragmatics, and phonology.
  Interventions: Behavioral: Conventional language intervention
- Developmental language disorder cases (Experimental): Developmental language disorder children who will receive the proposed narrative intervention program. The program will include 24 illustrated story sequences with a minimum of 5 sequences representing the main story elements: characters and setting; problems; internal response; actions; and consequence. Story icons will be designed to represent the main 5 elements to accompany storytelling and act as visual prompts.The narrative intervention program will be applied on the cases groups by a phoniatrician in 24 sessions, 60 minutes in duration, one session per week, for 3 months.
  Interventions: Behavioral: Narrative language intervention program
- Developmental language disorder control (Active Comparator): The developmental language disorder control group will receive the conventional language rehabilitation sessions in 30 minute sessions twice a week, for 3 months. Conventional language therapy targets semantics, syntax, prosody, pragmatics, and phonology.
  Interventions: Behavioral: Conventional language intervention

INTERVENTIONS:
Behavioral: Narrative language intervention program — Narrative language targets improving narrative macrostructure and microstructure.
  The program will include 24 illustrated story sequences with a minimum of 5 sequences representing the main story elements: characters and setting; problems; internal response; actions; and consequence. Story icons will be designed to represent the main 5 elements to accompany storytelling and act as visual prompts.
  Each story will reflect specific content with several target vocabulary words and complex morphosyntax. Each story will be followed by comprehension questions to facilitate understanding and answering question about stories.
  The following procedure will be implemented with each story: Modeling, answering comprehension questions, retelling with icons and colored illustrations, retelling with icons only, and retelling without icons. This procedure is adapted from story champs intervention program
  Arms: Developmental language disorder cases; Hearing Impairment cases
Behavioral: Conventional language intervention — Language rehabilitation targets improving semantics, syntax, pragmatics and phonology.
  Arms: Developmental language disorder control; Hearing Impairment control

SUMMARY:
The importance of narrative skills is evident in their role in language development and their relation to important academic skills namely reading, comprehension, and writing. Narratives are also essential for competent social skills, and children with delayed language development are usually found to have less proficient social communication skills. Research demonstrates the effects of narrative language intervention on improved narrative structure and complexity in addition to improved receptive and expressive use of syntax, morphology and general language use in children with narrative language impairment in various types of communication disorders. Given the importance of narrative language abilities in language development and due to lack of research targeting the assessment and intervention of narrative language skills of Arabic speaking children with language impairments, this study is dedicated towards the assessment of narrative language in Arabic speaking children and the development of a comprehensive intervention program targeting narrative language skills and its application on children with hearing impairment and developmental language disorder.

DETAILED DESCRIPTION:
A narrative refers to the ability to produce a fictional or real account of temporally sequenced meaningful occurrences and experiences. Studies have shown that narrative competence increases with age alongside language, cognitive and social skills. Development of narrative abilities starts during the preschool years, expands during the school age years, and continues to develop through adolescence and even adulthood.

Children with developmental language disorder (DLD) are known to have impaired narrative skills. Narratives of children with DLD are characterized by incomplete episodes, poor coherence, less expression of cognitive states, less complex sentences with fewer dependent clauses, and less complex morpho-syntax when compared to their peers.

Research has also shown that hearing impairment is another communication disorder in which narrative skills are particularly vulnerable. Narratives of children with hearing loss demonstrate comprehension and production deficits and they have a statistically significant lower performance in tests assessing narrative structure.

The aim of this work is to develop a narrative language intervention program and to apply it on children with developmental language disorder and children with hearing impairment to detect its efficacy on improving their narrative and language skills.

This study will be conducted on 44 children with hearing impairment, and 44 children with developmental language disorder attending the Unit of Phoniatrics, in the outpatient clinic of Alexandria Main University hospital. Sample size was calculated to achieve 80% power with a target significance level at 5% to detect the efficacy of the proposed narrative intervention program in improvement of narrative language skills of Egyptian children with hearing impairment and developmental language disorder.

The narrative intervention program will include an introductory section on the elements of story grammar to introduce the children to narratives and give them explicit instructions about the concepts of narrative macrostructure. The program will include 24 illustrated story sequences with a minimum of 5 sequences representing the main story elements: characters and setting; problems; internal response; actions; and consequence. Story icons will be designed to represent the main 5 elements to accompany storytelling and act as visual prompts. Each story will reflect specific content with several target vocabulary words and complex morphosyntax.

The following procedure will be implemented with each story: Modeling, answering comprehension questions, retelling with icons and colored illustrations, retelling with icons only, and retelling without icons.

All subjects meeting the specified inclusion and exclusion criteria will be assessed by the specified protocol of assessment to evaluate narrative skills, language skills and cognitive abilities before and after intervention.

The results of this study will be tabulated and analyzed with the use of appropriate statistical methods and appropriate figures and diagrams.

ELIGIBILITY:
Inclusion Criteria:

1. Children with developmental language disorder of both sexes in the age group (5 to 12 years).
2. Hearing-impaired children of both sexes with sensorineural hearing loss using auditory verbal communication in the age group (5 to 12) years with a minimum 2 years of experience with their hearing aids or cochlear implants with good benefit (hearing threshold less than 40 dB across all frequencies).
3. Hearing impaired children using hearing aids with pure tone average thresholds at 500, 1000, and 2000 Hz between 50 and 75 dB in unaided conditions.
4. Children with expressive language skills of at least 3 word length sentences.

Exclusion Criteria:

1. Children with intellectual disability.
2. Children with neurodevelopmental disorders (example; ASD).
3. Children with additional sensory deprivation (impaired vision).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-05-19 (Actual); Study Completion 2024-05-19 (Actual)

PRIMARY OUTCOMES:
Change in Test on Narrative language- second edition comprehension sub-test | baseline and 3 months
  The comprehension sub-test of the test of narrative language is a quantitative tol that assesses the ability to answer comprehension questions about 3 stories with a total maximum score of 47.
Change in Test on Narrative language- second edition production sub-test | baseline and 3 months
  The production sub-test of the test of narrative language is a quantitative tool that assesses the ability to tell 3 stories with a total maximum score of 88
Change in Test on Narrative language- second edition narrative language ability index | baseline and 3 months
  The comprehension and production subtests are combined to form a composite (narrative language ability index).

SECONDARY OUTCOMES:
change in comprehensive Arabic language test scores | baseline and 3 months
  Quantitative tool that evaluates language skills, raw scores are converted into language age equivalent scores
Change in values of Stanford Binet scale | baseline and 3 months
  Quantitative tool that evaluates verbal Intelligence, abstract intelligence and short term memory

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Ibrahim, Master, Principal Investigator — Alexandria University; Ossama A Sobhy, PhD, Study Chair — Alexandria University; Riham M ElMaghraby, PhD, Study Chair — Alexandria University; Nesrine H Hammouda, PhD, Study Director — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No